CLINICAL TRIAL: NCT07389304
Title: [EFFECTS OF SELECTED STATINS ON CARDIOVASCULAR PARAMETERS IN HEALTHY VOLUNTEERS: A RANDAMOZIED PHASE I CLINICAL TRIAL]
Brief Title: [Effects of Selected Statins on Cardiovascular Parameters in Healthy Volunteers]
Acronym: SBBU/IRC-25-31
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shaheed Benazir Bhutto University Sheringal Dir Upper (Other)
Collaborators: Khyber Medical University Peshawar (Other)
Responsible Party: Principal Investigator, Dr Abid Ullah, Lecturer, Shaheed Benazir Bhutto University Sheringal Dir Upper
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: [SBBU/PHM-25-32]; SBBU/IREC-25-32] (Other: [ShaheedBenazirBhuttoUSheringalDU])
Record Dates: First submitted 2026-01-20; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Lipid Profile,Blood Pressure
Keywords: sBlood Pressure,ECG change
MeSH Terms: interventions — Rosuvastatin Calcium; Atorvastatin; Simvastatin

STUDY DESIGN:
Intervention Model Description: The selected statins i.e Simvastatin (5mg, 20mg, 40mg), atorvastatin (10mg,20mg, 40mg) and simvastatin(10mg, 20mg, 40mg) will be given orally to the participants of different assigned randomized participants groups in once daily dosing for two days to assess the effect on blood pressure and ECG.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The PI will give the assigned medication to each participant according to randomization and allocation. All the personnel involved in the study will be kept blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rosuvastatin (5mg, 20mg, 40mg) (Experimental): The assigned participants will be given Rosuvastatin 5mg, 20mg, 40mg OD for two days
  Interventions: Drug: Rosuvastatin (5mg, 20mg, 40mg)
- Atorvastatin (10mg,20mg, 40mg) (Experimental): The assigned participants will be given Atorvastatin 10mg,20mg, 40mg OD for two days
  Interventions: Drug: Atorvastatin (10mg, 20mg, 40mg)
- Simvastatin (10mg, 20mg, 40mg) (Experimental): The assigned participants will be given Simvastatin 10mg, 20mg, 40mg OD for two days
  Interventions: Drug: Simvastatin (10mg, 20mg, 40m

INTERVENTIONS:
Drug: Rosuvastatin (5mg, 20mg, 40mg) — The Rosuvastatin (5mg, 20mg, 40mg) group participants will be given the drug orally OD for two days
  Arms: Rosuvastatin (5mg, 20mg, 40mg)
Drug: Atorvastatin (10mg, 20mg, 40mg) — The Atorvastatin (10mg, 20mg, 40mg) group participants will be given the drug orally OD for two days
  Arms: Atorvastatin (10mg,20mg, 40mg)
Drug: Simvastatin (10mg, 20mg, 40m — The Simvastatin (10mg, 20mg, 40mg) group participants will be given the drug orally OD for two days
  Arms: Simvastatin (10mg, 20mg, 40mg)

SUMMARY:
This study is a Phase I randomized clinical trial aiming to investigate the short-term effects of three commonly prescribed statins i.e (Atorvastatin, Rosuvastatin, and Simvastatin) at different dose levels i.e lo,median and high doses on cardiovascular parameters i.e Blood pressure and ECG morphology in healthy volunteers. The study will assess changes in blood pressure and ECG morphology following two days of statin administration under controlled conditions.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the effects of these three statins on the cardiovascular parameters in a dose-dependent manner. In this Phase 1 clinical trial we will enroll healthy volunteers who will be randomized to receive one of three statins at low, moderate, or high doses for two days. .

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Normal ECG
* Normal Blood Pressure
* Normal lipid levels

Exclusion Criteria:

* Participants with a history of diabetes mellitus,BP
* With chronic diseases e.g heart disease, kidney disease
* QTc ≥450 ms (men) or ≥470 ms (women)
* ECG changes
* Electrolyte imbalance,
* Participants taking other medications

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure Measurements | before dosing and 2 days after dosing achieving peak plasma concentrations respectively]
  Blood Pressure of the subjects will be determined by sphygmomanometer

SECONDARY OUTCOMES:
Electrocardiograms (ECGs) Measurements | before dosing and 2 days after dosing achieving peak plasma concentrations respectively]
  ECGs of the subjects will be determined by 12 Leads ECG Machine.QT interval and QRS complex in milliseconds will be analyzed to determine the effects of these statins on ECG morphology

CONTACTS AND LOCATIONS:
Locations (1):
- Shaheed Benazir Bhutto University Sheringal Dir Upper, Dīr, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The study results will be shared in well reputable Journals without the participant identifiers
Supporting Information: CSR